CLINICAL TRIAL: NCT06980961
Title: Short-pulse and Ultra-Short Pulse ND: YAG 1064 Lasers for Stasis Dermatitis Secondary to Chronic Venous Hypertension Treatment: the SUPERSTAR Trial
Brief Title: Short and Ultra-short-pulse ND: YAG 1064nm Lasers (Omer Smart and Omer Premium) for Stasis Dermatitis
Acronym: SUPERSTAR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Science Valley Research Institute (Other)
Responsible Party: Principal Investigator, Eduardo Ramacciotti, Senior investigator, Science Valley Research Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SUPERSTAR trial
Record Dates: First submitted 2025-04-30; First posted 2025-05-20 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Stasis Dermatitis
Keywords: laser; stasis dermatitis; hyperchromic skin lesions

STUDY DESIGN:
Intervention Model Description: 3 arms parallel study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1: ND YAG laser: 1064 nm short pulse (nanoseconds) - Omer Smart (Experimental): Laser treatment
  Interventions: Procedure: short-pulse ND: YAG 1064 laser
- Arm 2: ND YAG laser: 1064 nm ultra- short pulse (picoseconds) - omer Premium (Experimental): Laser treatment
  Interventions: Procedure: ultra-short-pulse ND: YAG 1064 laser
- Arm 3 (Placebo Comparator): Control vehicle (cold cream)
  Interventions: Drug: cold cream

INTERVENTIONS:
Procedure: short-pulse ND: YAG 1064 laser — Nd: YAG 1064 nm short pulse laser (5 nanoseconds), 4 mm spot size, from 100 to 1000 mJ total energy, treatment scheduled for six visits with pre-defined dates, with intervals of 28 to 35 days. The device will be Omer Smart, a Q-Switch Laser produced by Medical San (Lajeado, RS, Brazil).
  Other Names: Arm 1
  Arms: Arm 1: ND YAG laser: 1064 nm short pulse (nanoseconds) - Omer Smart
Procedure: ultra-short-pulse ND: YAG 1064 laser — Nd: YAG1064 nm ultra-short pulse laser (400 picoseconds), 2 to 10 mm spot size, from 100 to 1000 mJ total energy, treatment scheduled for 6 visits with pre-defined dates, with intervals of 28 to 35 days. The device will be Omer Premium, a picolaser produced by Medical San (Lajeado, RS, Brazil).
  Arms: Arm 2: ND YAG laser: 1064 nm ultra- short pulse (picoseconds) - omer Premium
Drug: cold cream — The control vehicle is a cold cream, supplied by HERVA'S manipulation pharmacy. The composition of cold cream will be beeswax, acetyl palmitate, BHA, cetearyl alcohol, propylparaben, and water. This topical agent will be applied to patients daily throughout the treatment period. It is scheduled for six visits with pre-defined dates, with intervals of 28 to 35 days.
  Arms: Arm 3

SUMMARY:
This study tests two types of lasers (ND YAG 1064 short and ultra-short pulses) to treat hyperchromic skin lesions secondary to venous hypertension (stasis dermatitis)

DETAILED DESCRIPTION:
Background: Stasis dermatitis with hyperpigmented skin lesions is a serious health problem for patients with chronic venous hypertension. Although no randomized studies have evaluated lasers for this treatment, lasers can be an attractive option.

Methods: This prospective, randomized, 3-arm, open-label, vehicle-controlled study will enroll patients scheduled to undergo treatment for stasis dermatitis with hyperpigmented skin lesions. Patients will be allocated to either Nd: YAG 1064 nm short pulse laser-nanoseconds (group 1), or Nd: YAG 1064 nm ultra-short-pulse laser-picoseconds (group 2), or cold cream vehicle control (group 3). All treatments are scheduled for 6 visits with pre-defined dates, with a final follow-up visit at intervals of 28 to 35 days. Primary outcomes include colorimetry analysis, secondary outcomes pre- and post-photographic analysis, and DLQI quality-of-life assessment.

Conclusions: The results of this trial will provide high-quality evidence to guide clinical practice on optimal management of hyperpigmented skin lesions secondary to stasis dermatitis.

ELIGIBILITY:
Inclusion Criteria:

1. Women or men aged 18 to 89 years with stasis dermatitis secondary to venous hypertension
2. Agreement with the terms of the survey and signing of the informed consent form
3. Availability to make the necessary appointments for treatment and follow-up
4. Provide consent to avoid pregnancy during treatment
5. Have primary venous hypertension already treated (treatment of varicose veins of the lower limbs) by any of the available techniques

Exclusion Criteria:

1. Men and women with CEAP 2 to 6, low mobility, no stasis dermatitis.
2. Peripheral arterial disease.
3. History of known allergy to the drugs used in this study
4. Presence of other types of dermatitis in the lower extremities, such as allergic stasis eczema.
5. Presence of comorbidities (such as diabetes mellitus, heart failure, respiratory failure, hypertension, hypothyroidism, or hyperthyroidism), pregnancy, breastfeeding, pulmonary hypertension, deep vein thrombosis (DVT), family history of DVT, known hypercoagulable states or thrombophilia, asthma, and migraine.
6. Anyone who does not agree with any of the search terms.

   -

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-05-20 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Colorimetry | 6 months
  The skin tone dissimilarity (expressed as ΔE) at treated and adjacent areas measured with digital calorimetry. The ΔE value derives from the differences in the International Commission on Illumination L*a*b* (CIELAB) color space. It is a structured approach to quantifying color differences, with specific intervals indicating varying levels of perceptibility with different intensities of pigmentation:
  * 0 < ∆E < 1 - the difference is unnoticeable
  * 1 < ∆E< 2 - the difference is only noticed by an experienced observer (mild),
  * 2 < ∆E < 3.5 - the difference is also noticed by an inexperienced observer (light),
  * 3.5 < ∆E < 5 - the difference is noticeable (moderate),
  * 5 < ∆E - gives the impression that these are two different colors (intense) In all sessions, patients will be submitted to colorimetric analysis. The ∆E is the skin color difference between the treated and adjacent areas.

SECONDARY OUTCOMES:
Photographic analysis | 6 months
  The co-primary outcome will be the incidence of post-procedure skin hyperpigmentation improvement after six treatment sessions, evaluated through before-and-after photo documentation analysis by three experienced, independent, and blind observers.
  All the evaluators will have access to high-definition before-and-after pictures of the patient's legs that were designated for them. Then, according to their expertise, they will answer the question, "Do you think there's post-treatment improvement in hyperpigmentation in the treated areas of this limb, yes or no?" for the affected limb. The answers chosen by most of the evaluators will be considered for data analysis.
Number of participants with treatment-related adverse events as assessed by clinical evaluation. | 6 months
  Safety analysis will be carried out by clinical evaluation in all pre-scheduled visits. It includes clinical analysis of potential skin alterations such as abnormal redness, swelling, temporary changes in skin pigmentation (hyper- or hypopigmentation), petechia, scarring, or burns. It will be reported as the number of participants with treatment-related adverse events.

OTHER OUTCOMES:
DLQI - quality-of-life | 6 months
  The DLQI will be applied in the baseline and final visits and includes 10 questions:
  1. Symptoms: How itchy, sore, painful, or stinging the skin has been.
  2. Embarrassment: How embarrassed or self-conscious one has been due to their skin.
  3. Daily Activities: How much has the skin condition interfered with shopping, home care, or gardening?
  4. Clothing: How much has the skin condition influenced the clothes worn?
  5. Social/Leisure: How much has the skin condition affected social or leisure activities?
  6. Sport: How much the skin condition has made it difficult to do sports.
  7. Work/Study: Whether the skin condition has prevented working or studying, and if not, how much it has been a problem.
  8. Personal Relationships: How much the skin condition has created problems with close relationships.
  9. Sex: How much the skin condition has caused sexual difficulties.
  10. Treatment: How much the treatment for the skin condition has been a problem, considering factors like time or mess.

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Ramacciotti, MD, Ph.D, livre docente, Study Chair — Science Valley Research Institute
Locations (1):
- Clinica Ramacciotti, Santo André, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Anonymized participant data can be made available upon requests directed to the corresponding author. Proposals will be reviewed based on scientific merit. After a proposal is approved, data can be shared through a secure online platform upon signing a data access agreement.
Supporting Information: Study Protocol, ICF
Time Frame: 2 years
Access Criteria: Anonymised participant data can be made available upon requests directed to the corresponding author. Proposals will be reviewed on the basis of scientific merit. After approval of a proposal, data can be shared through a secure online platform after signing a data access agreement.

REFERENCES:
- [Background] Vyas J, Johns JR, Ali FM, Ingram JR, Salek S, Finlay AY. A Systematic Review of 207 Studies Describing Validation Aspects of the Dermatology Life Quality Index. Acta Derm Venereol. 2024 Nov 7;104:adv41120. doi: 10.2340/actadv.v104.41120. PMID 39508500
- [Background] Liu C, Huang HY, Chang YY, Sun CK, Chia SH, Liao YH. Optical Effects of Focused Fractional Nanosecond 1064-nm Nd:YAG Laser: Techniques of Application on Human Skin. Lasers Surg Med. 2024 Aug;56(6):557-563. doi: 10.1002/lsm.23812. Epub 2024 Jun 18. PMID 38890780
- [Background] Ma S, Zhu H, Chen J, Chen F, Wu Y, He S, Li Y, Gong Y, Zhu H. Analysis of efficacy of picosecond laser treatment for nevus of Ota. Lasers Med Sci. 2025 Feb 6;40(1):72. doi: 10.1007/s10103-025-04322-0. PMID 39913065
- [Background] Silverberg JI, Kirsner RS, Margolis DJ, Tharp M, Myers DE, Annis K, Graham D, Zang C, Vlahos BL, Sanders P. Efficacy and safety of crisaborole ointment, 2%, in participants aged >/=45 years with stasis dermatitis: Results from a fully decentralized, randomized, proof-of-concept phase 2a study. J Am Acad Dermatol. 2024 May;90(5):945-952. doi: 10.1016/j.jaad.2023.12.048. Epub 2024 Feb 8. PMID 38340127
- [Background] Shriver MD, Parra EJ. Comparison of narrow-band reflectance spectroscopy and tristimulus colorimetry for measurements of skin and hair color in persons of different biological ancestry. Am J Phys Anthropol. 2000 May;112(1):17-27. doi: 10.1002/(SICI)1096-8644(200005)112:13.0.CO;2-D. PMID 10766940
- [Background] Basra MK, Chowdhury MM, Smith EV, Freemantle N, Piguet V. A review of the use of the dermatology life quality index as a criterion in clinical guidelines and health technology assessments in psoriasis and chronic hand eczema. Dermatol Clin. 2012 Apr;30(2):237-44, viii. doi: 10.1016/j.det.2011.11.002. Epub 2011 Dec 21. PMID 22284138
- [Background] Weatherall IL, Coombs BD. Skin color measurements in terms of CIELAB color space values. J Invest Dermatol. 1992 Oct;99(4):468-73. doi: 10.1111/1523-1747.ep12616156. PMID 1402005
- [Background] Ly BCK, Dyer EB, Feig JL, Chien AL, Del Bino S. Research Techniques Made Simple: Cutaneous Colorimetry: A Reliable Technique for Objective Skin Color Measurement. J Invest Dermatol. 2020 Jan;140(1):3-12.e1. doi: 10.1016/j.jid.2019.11.003. PMID 31864431
- [Background] Finlay AY, Khan GK. Dermatology Life Quality Index (DLQI)--a simple practical measure for routine clinical use. Clin Exp Dermatol. 1994 May;19(3):210-6. doi: 10.1111/j.1365-2230.1994.tb01167.x. PMID 8033378
- [Background] Liu J, Han C, Feng X, Liang J, Qu Y. Effective Picosecond Nd:YAG laser on seborrheic dermatitis and its mechanism. J Cosmet Dermatol. 2022 Jun;21(6):2449-2457. doi: 10.1111/jocd.14414. Epub 2021 Sep 8. PMID 34496116
- [Background] Eichenfield LF, Tom WL, Berger TG, Krol A, Paller AS, Schwarzenberger K, Bergman JN, Chamlin SL, Cohen DE, Cooper KD, Cordoro KM, Davis DM, Feldman SR, Hanifin JM, Margolis DJ, Silverman RA, Simpson EL, Williams HC, Elmets CA, Block J, Harrod CG, Smith Begolka W, Sidbury R. Guidelines of care for the management of atopic dermatitis: section 2. Management and treatment of atopic dermatitis with topical therapies. J Am Acad Dermatol. 2014 Jul;71(1):116-32. doi: 10.1016/j.jaad.2014.03.023. Epub 2014 May 9. PMID 24813302
- [Background] Dissemond J, Knab J, Lehnen M, Franckson T, Goos M. Successful treatment of stasis dermatitis with topical tacrolimus. Vasa. 2004 Nov;33(4):260-2. doi: 10.1024/0301-1526.33.4.260. PMID 15623206
- [Background] Silverberg JI, Hou A, Warshaw EM, Maibach HI, Belsito DV, DeKoven JG, Zug KA, Taylor JS, Sasseville D, Fransway AF, DeLeo VA, Pratt MD, Reeder MJ, Atwater AR, Fowler JF Jr, Zirwas MJ, Marks JG Jr. Prevalence and trend of allergen sensitization in patients with a diagnosis of stasis dermatitis referred for patch testing, North American contact dermatitis group data, 2001-2016. Arch Dermatol Res. 2022 Nov;314(9):857-867. doi: 10.1007/s00403-021-02295-y. Epub 2021 Nov 8. PMID 34748058
- [Background] Sundaresan S, Migden MR, Silapunt S. Stasis Dermatitis: Pathophysiology, Evaluation, and Management. Am J Clin Dermatol. 2017 Jun;18(3):383-390. doi: 10.1007/s40257-016-0250-0. PMID 28063094
- [Background] Abbade LP, Lastoria S, Rollo Hde A. Venous ulcer: clinical characteristics and risk factors. Int J Dermatol. 2011 Apr;50(4):405-11. doi: 10.1111/j.1365-4632.2010.04654.x. PMID 21413949
- [Background] Bergan JJ, Schmid-Schonbein GW, Smith PD, Nicolaides AN, Boisseau MR, Eklof B. Chronic venous disease. N Engl J Med. 2006 Aug 3;355(5):488-98. doi: 10.1056/NEJMra055289. No abstract available. PMID 16885552